CLINICAL TRIAL: NCT05474040
Title: Opioid-Sparing Multimodal Analgesia Versus Opioid Analgesia for Postoperative Pain After Elective Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, DR, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8099-12-10-2021
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Analgesia Post Craniotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid (Active Comparator): 2.5mg/iv morphine every 6hr postoperative
  Interventions: Drug: Morphine versus multimodal analgesia for post elective craniotomy pain
- multimodal (Active Comparator): combination of Gabapentin Orally (600 mg) the night before surgery and 2 hours before anesthesia induction plus dexmedetomidineIV bolus 1 μg/kg/10min + infusion pump 0.5 μg /kg/hrs intraoperative. Bupivacaine(scalp block) R/A 20ml 0.5% Postoperative. Acetaminophen IV 10-15 mg/kg 8hr postoperative. NSAIDs(ketorolac IV15-30mg every 6 postoperative
  Interventions: Drug: Morphine versus multimodal analgesia for post elective craniotomy pain

INTERVENTIONS:
Drug: Morphine versus multimodal analgesia for post elective craniotomy pain — To compare the effectiveness of opioid- sparing multimodal analgesia and opioid analgesia in the treatment of post-craniotomy pain

SUMMARY:
Several neurosurgical procedures can cause postoperative pain including craniotomies for tumor resections, epilepsy surgery and craniotomies for aneurysm clipping, penetrating traumatic brain injury, and neuroradiological procedures such as arteriovenous embolization procedures and aneurysm coiling's. Postoperative hematomas, elevation of intracranial pressures, cerebral infarctions, seizures, hypertension, development of air embolism, cranial nerve injury, and the development of cerebral edema and stroke can complicate the management of postoperative pain .

Within the initial 24 hours post craniotomy, 60% of patients experienced moderate-to-severe pain. Most patients describe the pain as predominantly superficial suggesting a pathogenesis that is somatic instead of visceral. It is believed to originate from soft tissue and per cranial muscle, rather than the brain tissue itself .

Majority of patients undergoing craniotomy experienced severe pain in surgical site after the procedure.Insufficient pain control after craniotomy can increase the intracranial pressure in patients with compromised cerebral auto regulation, and arterial or intracranial hypertension can lead to intracranial hemorrhage .

Moreover, most neurosurgeons want to ascertain the neurological results as early as possible, so cautious postoperative pain management is required so as not to disturb the neurological assessment after craniotomy .

As a consequence of these conflicting scenarios and emerging interest in avoiding opioids, there is greater emphasis on sparing -opioid alternatives, as well as growing interest in the use of opioid-free anesthesia and perioperative analgesia .

If the need for opiates is eliminated for these patient it will improve post-operative neurological examination significantly and hopefully decrease the number of investigations (e.g. computed tomography [CT] scans) due to more reliable clinical examination .

There is lack of consensus and evidence regarding the use of common systemic analgesics for post craniotomy pain. Analgesic adjuvants like Paracetamol, NSAIDs, gabapentin, dexmedetomedine, scalp block can be used alone or in combination. When various analgesic drugs of different classes, different mechanisms of action, and adverse-effect profiles are used in combination, this may result in synergism of the analgesic effects. This method is called Multimodal analgesia, it is considered very effective and optimum for management of post craniotomy pain, in addition to opioid sparing effect .

Rationale Stress response to pain after craniotomy procedure in the form of hemodynamic changes (hypertension and tachycardia) and increase in intracranial tension, can cause serious intracranial complications.Opioids are the most commonly used agents for treating moderate to severe postoperative pain, however it usually associated with adverse effects such as postoperative nausea and vomiting, respiratory depression and excessive sedation.Previous studies showed that combined use of multimodal opioid sparing analgesics such as Paracetamol, NSAIDs, Gabapentin, Dexamdetomedine, scalp block offers the promise of improved pain and reduced opioid consumption while preserving the clinical neurologic examination. Research question: Is multimodal opioid sparing analgesia safer, beneficial and more effective than opioids for post craniotomy analgesia? Aim of the study Adequate analgesia with less opioid consumption and related side effects in patients with elective craniotomy.

Objectives

1. To compare the effectiveness of opioid- sparing and opioid analgesia in the treatment of post-craniotomy pain: regarding pain relief time to the first rescue analgesia and total dose of postoperative analgesia.
2. To compare adverse effects between opioid and opioid- sparing analgesia groups such as postoperative nausea and vomiting and excessive sedation.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patient consent. 2. Age : (21 to 65) years. 3. Sex : both. 4. ASA grade I-II (American society of anesthiologists). 5. Prepared to elective craniotomy under general anesthesia (for eg draining of Abscess, tumor, blood clot or aneurysm).

6. Ability to take pills

Exclusion Criteria:

* 1. Disturbed conscious level (Glascow coma score less than14). 2. Previous craniotomy. 3. Chronic use of analgesics or drug dependence or regular anticonvulsant, neuropathic or antidepressant use.

  4. Uncontrolled hypertension. 5. Extensive surgeries lasting more than 6 hours or patient needing postoperative ventilator support.

  6. Intracranial malformations. 7. Any complications during procedure such as massive intracranial hemorrhage. 8. Psychological disorder requiring pharmacologic treatment. 9. Regular systemic steroid use. 10. Renal impairment or liver dysfunction. 11. Allergy 12. Bleeding tendency

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
pain score by VAS | 24 hours
  To compare the effectiveness of opioid- sparing and opioid analgesia in the treatment of post-craniotomy pain

SECONDARY OUTCOMES:
post medications complications | 24 hours
  To compare adverse effects between opioid and opioid- sparing analgesia groups such as postoperative nausea and vomiting and excessive sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Essamedin Negm, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided